CLINICAL TRIAL: NCT04249726
Title: The Restoration of Minimally Destructed Posterior Endodontically Treated Teeth Using Indirect Full Coverage Restorations Compared to Direct Composite Resin Restorations: A Randomised Clinical Trial.
Brief Title: The Restoration of Endodontically Treated Teeth Using Indirect Full Coverage Restorations Compared to Direct Composite Resin Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Motasum Abu-Awwad, Assistant Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UJordan1
Record Dates: First submitted 2020-01-24; First posted 2020-01-31 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Intervention Model Description: Two groups parallel to each other randomly assigned to a specific intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct composite resin restoration (Experimental): Root filled teeth with occlusal cavities and at least 3 intact axial walls will receive composite resin restorations
  Interventions: Procedure: Direct composite resin restoration
- Full coverage metal-ceramic crown (Active Comparator): Root filled teeth with occlusal cavities and at least 3 intact axial walls will receive composite resin restorations followed by full coverage metal-ceramic crown
  Interventions: Procedure: Direct composite resin restoration followed by full coverage metal ceramic crown

INTERVENTIONS:
Procedure: Direct composite resin restoration — A direct composite resin restoration will be provided intracoronally without cuspal coverage.
  Other Names: Intracoronal restoration
  Arms: Direct composite resin restoration
Procedure: Direct composite resin restoration followed by full coverage metal ceramic crown — A direct composite resin restoration will be provided intracoronally followed by a full cuspal coverage metal ceramic crown.
  Other Names: Full coverage metal-ceramic crown
  Arms: Full coverage metal-ceramic crown

SUMMARY:
The use of full cuspal coverage restoration for the management root treated teeth was advocated by many clinical studies and supported by systematic reviews. However, most of the studies did not take into account the amount of tooth structure remaining before providing cuspal coverage. The strength and fracture resistance of the tooth has been shown to be positively correlated with the amount of tooth structure remaining. A more conservative treatment option could be selected for a root treated tooth with good amount of remaining tooth structure such as direct restorations.

The aims of this randomized clinical trial is to compare the survival and success of root treated teeth with occlusal cavities and at least three intact axial walls, when restored through the use of indirect full cuspal coverage restorations vs direct composite resin restorations.

DETAILED DESCRIPTION:
The management of posterior endodontically treated teeth (ETT) is still to this day considered a controversial topic.The use of full cuspal coverage restoration for the management ETT was advocated by many clinical studies and supported by systematic reviews. However, most of the studies did not take into account the amount of tooth structure remaining before providing cuspal coverage. An ETT tooth with an MOD cavity will be at a higher risk of fracture than an ETT tooth with just an occlusal cavity. Managing both with cuspal coverage could be considered an overtreatment and an unnecessary removal of tooth structure. The strength and fracture resistance of the tooth has been shown to be positively correlated with the amount of tooth structure remaining. A more conservative treatment option could be selected for an ETT with good amount of remaining tooth structure such as direct restorations.

The aims of this randomized clinical trial is to compare the survival and success of ETT with occlusal cavities and at least three intact axial walls, when restored through the use of indirect full cuspal coverage restorations vs direct composite resin restorations.

The groups are:

Group 1: Managed with direct intracoronal composite resin restoration. Group 2: Managed with a direct composite resin restoration, followed by an indirect full coverage restoration.

Patients will be recalled at 1 year, 3 years and 5 years.

Treatment protocol for each group Group 1: Patient receiving a composite resin restoration. Following rubber dam isolation, the temporary restoration will be removed. The enamel will be selectively etched with 37% phosphoric acid and rinsed and dried thoroughly till a white frost appearance appeared. An adhesive system (ScotchBond Multi-Purpose - 3M ESPE) will then be applied to the dentine according to the manufacturer instructions and then will be cured for 30 seconds. The direct restoration will be made using a microhybrid resin composite (Filtek Z350, 3M ESPE), which will be applied in increments and each increment cured for 40 seconds. Glycerin will be applied to the final restoration and cured for 5 seconds to prevent the development of the oxygen inhibition layer. The restoration will then be finished with ultra-fine diamond finishing burs, and polished with Sof-Lex discs (3M ESPE) and 0.1 micrometer particle size diamond paste. Occlusion will be checked to conform to the patient's current occlusion status and make sure no interferences were introduced.

Group 2: Patients receiving a composite resin restoration and followed with an indirect full coverage restoration.

The same steps used as for group 1 would be followed to build the composite resin core. This will be followed with a preparation for the indirect full cuspal restoration. Three additional silicone putty indices will be made; one will be made for the production of a provisional crown, and the other two will be cut and used as reduction indices (one will be cut mesio-distally and the other one will be cut facially-lingually/palatally). The preparation will be carried out with diamond burs. The guidelines to be followed will include:

* Supra or equigingival margins if aesthetic was of concern.
* Chamfer finish-line
* 2 mm occlusal reduction;
* 1.5 mm axial reduction all around Following the application of two double retraction cord sizes 00 and 0 (Ultradent), the impression will be made with additional silicone (Zermack) and the cast poured in Die stone. The crown will be fabricated in the laboratory.

The temporary crown made from self-cure bisacrylic (Protemp, 3M ESPE) would be cemented using Eugenol free temporary crown and bridge cement (TempBond). All crowns will be cemented after 1 week using Resin modified glass ionomer cement (RelyX luting plus, 3M ESPE).

Follow-up appointments and data Collection

Clinical evaluation will include:

* Visual inspection conducted with loops at magnification 4.5
* Examination of the continuity of the margins of the restoration with the tooth structure by use of an explorer
* Periodontal probing performed with a periodontal probe.
* Color photos (1:1 mirror shots) of the restorations were taken with standard film
* Periapical and bitewing radiographic examination was performed by use of a paralleling technique at 65 kV and 8 mA.
* Patients reported outcome measures (PROM)

Evaluation of success or failure will be performed by 2 examiners other than the operator.

ELIGIBILITY:
Inclusion Criteria:

* To have at least one posterior tooth in need for root canal treatment and restoration.
* The tooth structure loss of the tooth should be limited to an occlusal cavity with at least three remaining axial walls (>2mm thickness).
* The tooth should be opposed by a natural tooth or a fixed partial denture.
* The tooth should not be serving as an abutment for a removal or fixed partial denture.

Exclusion Criteria:

- Patients under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Survival | 5 years
  Survival of the tooth and restoration
Success | 5 years
  Success of the restoration without complications: to be assessed based on modified USPHS criteria (margin integrity, color, surface texture)
Complications | 5 years
  Complications that affect the restoration
Patient reported satisfaction | 5 years
  Patients' reported satisfaction with the restoration provided regarding: appearance, function, ease of cleaning and cost using the visual analog scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Jordan Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided